CLINICAL TRIAL: NCT00564317
Title: KIDNET vs Meditation/Relaxation - a Dissemination Randomized Controlled Trial for the Treatment of Traumatized Children After War in Sri Lanka
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: NGO vivo e.V. (Unknown); GTZ-German Technical Cooperation, Germany (Unknown); European Refugee Fund (Other); German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mb/19.10.05
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Post-Traumatic Stress Disorders
Keywords: PTSD; Depression; Suicidality; trauma-focussed treatment; KIDNET; Narrative Exposure Therapy for Children; Meditation; Relaxation; War
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Suicidal Ideation | interventions — Meditation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 KIDNET (Experimental): Narrative Exposure Therapy for Children
  Interventions: Behavioral: KIDNET
- 2 Meditation/Relaxation (Experimental): mixed Meditation/Relaxation Protocol
  Interventions: Behavioral: Meditation/Relaxation
- 3 KIDNET + Meditation/Relaxation (Experimental): KIDNET according to protocol, waiting time of 5 months, then Meditation/Relaxation according to protocol
  Interventions: Behavioral: KIDNET; Behavioral: Meditation/Relaxation
- 4 Meditation/Relaxation + KIDNET (Experimental): Med/Relax according to protocol, 5 months waiting time, KIDNET according to protocol
  Interventions: Behavioral: KIDNET; Behavioral: Meditation/Relaxation

INTERVENTIONS:
Behavioral: KIDNET — Narrative Exposure Therapy for Children - a short term intervention for the treatment of trauma after war, organized violence, torture, abuse and other detrimental life events
  Arms: 1 KIDNET; 3 KIDNET + Meditation/Relaxation; 4 Meditation/Relaxation + KIDNET
Behavioral: Meditation/Relaxation — a protocol of traditional/local meditation and relaxation exercises, such as breathing meditation, chanting, body relaxation
  Arms: 2 Meditation/Relaxation; 3 KIDNET + Meditation/Relaxation; 4 Meditation/Relaxation + KIDNET

SUMMARY:
The purpose of this study is to assess the efficacy of KIDNET versus a Meditation/Relaxation protocol in treating traumatized children when applied by locally trained teacher counsellors as well as the effectiveness and adequacy of such a treatment in a south-asian war affected stayee child community.

DETAILED DESCRIPTION:
Outcome measures include PTSD symptom score, Depression score, Suicidal ideation and related functioning measures (including school grades)

ELIGIBILITY:
Inclusion Criteria:

* all children with PTSD Diagnosis from six surveyed schools in Vallikamam/Jaffna educational zones age range 11-15

Exclusion Criteria:

* none

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2004-09; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
PTSD-Symptoms according to CAPS-CA (DSM-IV) | pre-test, 5-months, 14-months

SECONDARY OUTCOMES:
Depression score & Suicidality according to M.I.N.I. KID A and B | pre-test, 5-months, 14-months

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Rockstroh, Prof Dr, Principal Investigator — University of Konstanz; Elisabeth Schauer, MA/MPH, Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz/vivo e.V. Germany & Vallikamam/Jaffna Educational Zones, Sri Lanka, Jaffna/Vallikamam, Sri Lanka

REFERENCES:
- See also: website of NGO which supported implementation in the field — http://www.vivo.org